CLINICAL TRIAL: NCT03197012
Title: Yttrium-90 DOTA-TOC Intra-arterial (IA) Peptide Receptor Radionuclide Therapy (PRRT) for Neuroendocrine Tumor
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Thomas Hope (Other)
Responsible Party: Sponsor-Investigator, Thomas Hope, Assistant Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17455; NCI-2017-01886 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Neuroendocrine Tumor
Keywords: neuroendocrine tumor (NET); Peptide Receptor Radionuclide Therapy (PRRT); somatostatin receptor (SSTR)
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — 90Y-octreotide, DOTA-Tyr(3)-; gallium Ga 68 dotatate; Ga(III)-DOTATOC

STUDY DESIGN:
Intervention Model Description: Main study: All participants will receive a single administration of intra-arterial 90Y-DOTA-TOC.
  There will be a sub-study involving 10 patients from the main study who will undergo additionally correlative imaging to compare IA vs IV administration (intra-arterial 68Ga-DOTA-TOC administration and subsequent PET imaging).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Main Study: 90Y-DOTA-TOC (Experimental): 90Y-DOTA-TOC will be administered one time over thirty minutes via the hepatic arterial catheter in the outpatient setting. The injected dose will be 85 to 115 mCi.
  Interventions: Drug: 90Y-DOTA-TOC
- Sub-study: 90Y and 68Ga-DOTA-TOC (Experimental): 90Y-DOTA-TOC will be administered one time over thirty minutes via the hepatic arterial catheter in the outpatient setting. The injected dose will be 85 to 115 mCi.
  Patients enrolled in the correlative sub-study will also receive 111-259 MBq (3-7 mCi) of 68Ga-DOTA-TOC concurrent with 90Y-DOTA-TOC
  Interventions: Drug: 90Y-DOTA-TOC; Drug: 68Ga-DOTA-TOC

INTERVENTIONS:
Drug: 90Y-DOTA-TOC — Starting 30 minutes prior to the administration of 90Y-DOTA-TOC, amino acid solution will be administered via IV, and will continue through the PRRT procedure. An angiographic catheter will be inserted under fluoroscopic guidance to the appropriate location in the hepatic artery. 90Y-DOTA-TOC will be administered via the hepatic arterial catheter.
  Other Names: Yttrium-90 DOTATOC
Drug: 68Ga-DOTA-TOC — In the sub-study, 10 patients will receive 68Ga-DOTA-TOC concurrent with the 90Y-DOTA-TOC dose and 90 minutes after treatment, these patients will be imaged using a PET/CT. The following day, patients enrolled in the sub-study will undergo a PET/MRI.
  Other Names: Gallium-68 DOTATOC
  Arms: Sub-study: 90Y and 68Ga-DOTA-TOC

SUMMARY:
This is a prospective, pilot, single center, open-label study in patients with metastatic neuroendocrine tumor. Eligible participants will undergo baseline assessments at enrollment. Study participants will receive a one-time administration of 90Y-DOTA-TOC via the hepatic artery.

Participants in the correlative sub-study will receive 68Ga-DOTA-TOC concurrent with the 90Y-DOTA-TOC dose, and undergo additional imaging and assessment.

DETAILED DESCRIPTION:
Prior to the procedure, the patient will be instructed to fast overnight. Upon arrival to the hospital intravenous (IV) access will be placed, and Additionally, a scopolamine patch may be placed the night prior to treatment. Additionally a Foley catheter will be placed.

Starting 30 minutes prior to the administration of 90Y-DOTA-TOC, an amino acid solution will be administered via IV. An angiographic catheter will be directed under fluoroscopic guidance to the appropriate location in the hepatic artery.

The 90Y-DOTA-TOC dose will be administered over thirty minutes via the hepatic arterial catheter in an outpatient setting.

Ten patients also enrolled in the correlative sub-study will receive 68Ga-DOTA-TOC concurrent with the therapeutic dose and 90 minutes after treatment, these patients will be imaged 90 minutes after treatment using a Positron Emission Tomography (PET) combined with Computerized tomography (CT) (PET/CT) and the following day using Positron Emission Tomography (PET) combined with magnetic resonance imaging (MRI) (PET/MR).

All study participants will be followed up on protocol for six months for evaluation of toxicity and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven neuroendocrine tumor, which is somatostatin receptor positive as demonstrated on somatostatin receptor Positron Emission Tomography (PET).

1. All sites or origin are eligible.
2. Functional and nonfunctional tumors are allowed. 2. Hepatic metastases on imaging meeting the following criteria:

a. Liver-only or liver-dominant metastases, defined as: i. At least 10% liver parenchyma replacement by tumor, but less than 70% replacement of the hepatic parenchyma by tumor.

1. For the imaging sub-study: at least one liver lesion must measure greater than 2 cm in size 2. For the imaging sub-study: treatment must only be performed using a single dose, and so arterial variant anatomy that would result in a split treatment will not be allowed ii. And, progression of the liver metastases demonstrated within the past twelve months defined as either:

1. Appearance of any new liver lesion or
2. 20% increase in size of at least one liver lesion. iii. Presence of low-volume extrahepatic lesions (including primary tumor) is allowed if they are stable and asymptomatic.

   b. SUVmax on 68Ga-DOTA-TOC PET of the liver metastases two times greater than the adjacent liver parenchyma.
3. Not a candidate for surgical debulking.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
5. Age > 18.
6. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Patients not capable of getting PET study due to weight, claustrophobia, or inability to lie still for the duration of the exam.

   a. For patients in the imaging correlate sub-study: contraindication for undergoing MRI based on University of California, San Francisco (UCSF) Radiology guidelines.
2. Contraindication to hepatic arteriography (e.g. hepatic artery dissection and/or thrombosis, uncorrectable coagulopathy, severe allergy to iodinated contrast, severe vascular disease precluding safe hepatic artery catheterization).
3. Any patient receiving treatment with short-acting octreotide, which cannot be interrupted for 48 hours before and 24 hours after the administration of 90Y-DOTA-TOC, or any patient receiving treatment with octreotide long-acting release (LAR) or lanreotide, which cannot be interrupted for at least 4 weeks before the administration of 90Y-DOTA-TOC.

   a. Concurrent somatostatin receptor analog (SSA) allowed if progression has been documented and the SSA dose has been stable for at least two months. Long-acting SSA cannot be given within four weeks of treatment and short-acting SSA cannot be given with 48 hours of treatment. SSA therapy can restart one day after treatment.
4. Interferon, everolimus (mTOR-inhibitors), sunitinib or other systemic therapies within 4 weeks prior to enrollment. Bevacizumab within 6 weeks prior to enrollment.
5. Any liver directed treatment (surgery, radioembolization, chemoembolization, chemotherapy and radiofrequency ablation) within 12 weeks prior to enrollment.
6. Any external beam radiation treatment for hepatic disease. Prior external beam radiation therapy to more than 25% of the bone marrow.

   a. Prior systemic PRRT treatment is allowed, if it was performed at least six months prior.
7. Pregnancy or lactation. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation
8. Impaired liver function

   1. aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) / alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase (SGPT)) > 3 x upper limit of normal (ULN).
   2. Total bilirubin >1.5 x ULN
   3. Serum albumin <3.0 g/dL unless prothrombin time is within the normal range.
   4. Thrombosis of the main portal vein
   5. Clinical evidence of ascites (trace ascites on imaging acceptable).
9. Impaired bone marrow reserve

   1. Hb concentration < 8.0 g/dL;
   2. Total White Blood Cell count (WBC) <2x109/L (2000/mm3);
   3. Platelets <75x109/L (75x103/mm3).
10. Creatinine clearance <50 mL/min calculated by the Cockroft Gault method.
11. Known intracranial metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Over the duration of the study, which is estimated to be approximately 36 months
  Based on change in size of hepatic lesions three and six months after treatment with IA 90Y-DOTA-TOC using RECIST criteria.
Incidence of Treatment-Related Adverse Events [Safety] | Over the duration of the study, which is estimated to be approximately 36 months
  Based on laboratory evaluation and CTCAE 4.0 criteria.

SECONDARY OUTCOMES:
Change in SUVmax between pre-treatment IV 68Ga-DOTA-TOC PET and treatment IA 68Ga-DOTA-TOC. | Over the duration of the study, which is estimated to be approximately 36 months
  Data from patients in the imaging correlate sub-study only
Correlation between uptake on IA 68Ga-DOTA-TOC PET/CT compared to 24-hour post-treatment IA 90Y-DOTA-TOC PET/MRI. | Over the duration of the study, which is estimated to be approximately 36 months
  Data from patients in the imaging correlate sub-study only

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT03197012/ICF_000.pdf